CLINICAL TRIAL: NCT01878565
Title: The Treatment With Nucleoside Analogues in Combination With HBIG+GM-CSF+HBV Vaccine for Chronic Hepatitis B Patients With HBeAg Seroconversion: a Phase I/II, Single-blind, Randomized, GM-CSF-controlled Trial
Brief Title: The Treatment With HBIG+GM-CSF+HBV Vaccine for Chronic Hepatitis B Patients With HBeAg Seroconversion
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Principal Investigator, Fu-Sheng Wang, Research Center for Biotherapy, Beijing 302 Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Beijing302-009; yes (Other: Beijing 302 Hospital)
Record Dates: First submitted 2013-06-12; First posted 2013-06-17 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-07

CONDITIONS: Chronic Hepatitis B
Keywords: HBIg; GM-CSF; HBV vaccine; immune regulatory therapy
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Pharmaceutical Preparations; Drug and Narcotic Control

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug treatment (Experimental): Drug: Given four times in week 0, 4, 12 and 24. At each time of treatment, the patients will be hospitalized and treated with 800 unit of HBIG intramuscularly at day 0, 1, 2, 3 and 4, then were treated with 75 μg of GM-CSF subcutaneously at day 2, 3, 4, 5 and 6, and finally were injected 20μg of HBV vaccine subcutaneously at day 6.
  Interventions: Drug: Drug
- GM-CSF control (Other): GM-CSF was given four times as control in week 0, 4, 12 and 24. At each time of treatment, the patients will be hospitalized and treated with GM-CSF intramuscularly or subcutaneously at day 2, 3, 4, 5, 6.
  Interventions: Drug: GM-CSF control

INTERVENTIONS:
Drug: Drug — Given four times in week 0, 4, 12 and 24. At each time of treatment, the patients will be hospitalized and treated with 800 unit of HBIG intramuscularly at day 0, 1, 2, 3 and 4, then were treated with 75 μg of GM-CSF subcutaneously at day 2, 3, 4, 5 and 6, and finally were injected 20 μg of HBV vaccine subcutaneously at day 6.
  Other Names: treatment group
  Arms: Drug treatment
Drug: GM-CSF control — Given four times in week 0, 4, 12 and 24. At each time of treatment, the patients will be hospitalized and treated with saline placebo intramuscularly or subcutaneously at day 2, 3, 4, 5, 6.
  Other Names: drug control
  Arms: GM-CSF control

SUMMARY:
The host immunity has been generally recognized as the main factors to determine the outcome of chronic hepatitis B virus (HBV) infection; however, previous studies have shown that HBV-specific T cell and B cell function are exhausted in chronic hepatitis B (CHB) patients. Recently, It is suggested that hepatitis B surface antigen (HBsAg) may play a key role in the immune tolerance or immune exhaustion. Anti-HBV immune responses are partially recovered when patients achieved hepatitis B e antigen (HBeAg) seroconversion during antiviral therapy, and can be nearly recovered during HBsAg seroconversion. However, it is still difficult to achieve the ideal terminal, HBsAg seroconversion. For this reason, immunotherapy would be helpful to enhance the anti-HBV immunity and acquire higher HBsAg seroconversion. Here, the investigators propose a hypothesis that hepatitis B immune globin (HBIG)+granulocyte-macrophage colony-stimulating factor (GM-CSF)+HBV vaccine can enhance anti-HBV immune responses and improve HBsAg seroconversion in CHB patients who has achieved HBeAg seroconversion using nucleoside analogues treatment.

DETAILED DESCRIPTION:
The host immunity has been generally recognized as the main factors to determine the outcome of chronic hepatitis B virus (HBV) infection. Previous studies have shown that HBV-specific T cell and B cell function are exhausted in chronic hepatitis B (CHB) patients. Interestingly, these impaired T and B cell functions could be partially restored by antiviral treatment, but this recovery seemed to be uncompleted even if long-term HBV suppression and HBeAg seroconversion. Recently, several emerging evidences have indicated that HBV-specific immune responses could be nearly recovered after hepatitis B surface antigen (HBsAg) seroconversion. This phenomenon suggest that HBsAg may play a key role in the immune tolerance or immune exhaustion. Indeed, our recent studies have found that the patients with HBsAg seroconversion display an HBV-specific T and B cell responses. Thus, the amount of HBsAg may serve as a possible mechanism for evading the host immune response, while anti-HBs antibody and HBV specific-T cell responses provide protective immunity.

HBsAg was the Nobel prize discovery that identified HBV about 40 years ago; to this day HBsAg remains the hallmark of overt HBV infection. HBsAg synthesis during the HBV viral life cycle is complex, and typically occurs at the endoplasmic reticulum. The envelope open reading frame (ORF) contains pre-surface 1 (preS1), pre-surface 2 (preS2), and ORF-S domains and envelope proteins are generated from two HBV messenger ribonucleic acid (mRNA) transcripts, with subsequent translation resulting in small (ORF-S), medium (pres2 + ORF-S) and large surface envelope proteins (preS1 + preS2 + ORF-S). These are also known as large (L), medium (M) and small (S) surface proteins, respectively. However, HBsAg production far exceeds that required for virion assembly, and excess surface envelope proteins are secreted as non infectious filamentous or spherical sub-viral particles, which exceed virions by a variable factor of 102-105 and can accumulate up to concentrations of several hundred micrograms per milliliter of serum. These data suggested that sAg mainly derive from sub-viral particles, and the decline of serum HBsAg means reduction of covalently closed circular DNA (cccDNA) transcription and mRNA translation but not HBV replication. Recently, several studies suggest a new potential role of quantitative serum HBsAg in the prediction of virological response to antiviral therapy, at least in pegylated interferon (Peg-IFN) treated patients. In natural history of chronic HBV infection, HBsAg levels differ significantly during the 4 phases of HBV infection and decline progressively from immune tolerance (IT) (5 log IU/ml) to low replication (LC) (3 log IU/ml), while HBsAg/HBV-DNA ratios are significantly higher in LC as compared to all the others patients. These data suggested that the quantitative HBsAg may be a promising prognostic marker during the natural history of HBV-infection and during antiviral therapy. Thus, the loss of HBsAg and the development of anti-HBs antibodies (HBsAg-seroconversion) is the ultimate goal of anti-HBV therapy.

CHB patients would achieve HBV DNA replication inhibition, glutamic-pyruvic transaminase (ALT) normalization and hepatitis B e antigen (HBeAg) seroconversion after treatment with antiviral therapy. In addition, the antiviral immunity would be improved during the this process. However, it is difficult for these patients to clear HBsAg and reach the idea terminal. The major reasons are the presence of HBsAg and HBV-specific immunity was impaired. For this reason, immunotherapy would be helpful to enhance the anti-HBV immunity and acquire higher HBsAg seroconversion rate. The purpose of this study is to investigate whether and how immunotherapy ie. HBIG+GM-CSF+HBV vaccine improve the rate of HBsAg seroconversion. This study will also focus on the tolerance and safety of this treatment in CHB patients.

Participants in this study will be randomly assigned to one of two treatment arms:

Arm A: Participants will receive 48 weeks of nucleoside analogs (NAs) treatment combined with 24-week treatment with hepatitis B immune globin (HBIG)+granulocyte-macrophage colony-stimulating factor (GM-CSF)+HBV vaccine.

Arm B: Participants will receive 48 weeks of NAs treatment combined with 24-week treatment with saline placebo.

All of patients will be treated continuously with NAs for 48 weeks in combination with HBIg+GM-CSF+HBV vaccine treatment or saline placebo for first 24-week and then followed-up for other 24-week. In treatment period (24 weeks), the treatment of HBIg+GM-CSF+HBV vaccine will be given four times in week 0, 4, 12 and 24. At each time of treatment, the patients will be hospitalized and treated with 800 unit of HBIG intramuscularly at day 0, 1, 2, 3 and 4, and were treated with 75 μg of GM-CSF subcutaneously at day 2, 3, 4, 5 and 6, and finally were injected 20μg of HBV vaccine subcutaneously at day 6. This approach allow that the initial HBIG injection possibly reduces HBsAg, then antigen-presenting cells are activated by GM-CSF treatment, and finally HBV vaccine is used to priming APC to induce HBV-specific immune responses. In control group, the patients will received GM-CSF as control at each time. After treatment has been initialized, the participants will be asked to come to the clinic on weeks 4, 12, 24, 36 and 48. At each visit participants will receive enough study treatment to last until the next visit. Each visit will last between 2 and 3 hours. At most visits participants will have a physical exam, answer questions about any medications they are taking and how they are feeling, and have blood drawn for safety and efficacy and HBsAg quantization. Some additional blood will also be stored for HBV-specific T cell and B cell responses. At some visits participants will be asked questions about their medication and medical history, have pupils dilated, have a hearing test, and have an electrocardiogram (EKG). Some visits will require participants to arrive fasting. Pregnancy tests may also be conducted so as to avoid some participants who is able to become pregnant or if pregnancy is suspected.

ELIGIBILITY:
Inclusion Criteria:

1. chronic hepatitis B patients with HBeAg seroconversion (eAg negative and eab positive)
2. age 18-50, male or female
3. HBsAg positive for at least 6 months, quantitative HBsAg <1000 IU/ml (Abbott Diagnostic, Wiesbaden, Germany)
4. HBeAg positive CHB patients who have received NAs (lamivudine, adefovir dipivoxil, entecavir, alone or in combination) treatment and achieved HBeAg seroconversion (HBeAg-, HBeAb+), HBV DNA<40 IU/ml and ALT normalization and maintained for at least 6 months.
5. Urine pregnancy test is negative in gestational age female subjects before enrollment, who can take effective contraceptive measures and agree to contraception during treatment and follow-up period.
6. Enrolled subjects should understand and sign the informed consent and comply with the requirement of the research before study.
7. Enrolled subjects should agree not to participate in other studies, and not to accept other immunomodulatory therapy during the study. Other treatments such as corticosteroids should be informed timely

Exclusion Criteria:

1. Be allergic to HBIG, GM-CSF and HBV vaccine.
2. Coinfected with other virus. Any positive for anti-hepatitis A virus (HAV), anti-hepatitis C virus (HCV), anti-hepatitis D virus (HDV), anti-hepatitis E virus (HEV) and anti-HIV.
3. Advanced cirrhosis or Child-Pugh 7 scores or above.
4. Autoimmune thrombocytopenic purpura, coronary heart disease, cerebrovascular disease, hypertension, diabetes mellitus, high myopia, history of epilepsy.
5. Other causes of liver disease, such as autoimmune liver disease, alcoholic liver disease, nonalcoholic liver disease, drug-induced liver disease and other unknown causes of chronic liver diseases.
6. Associated with other serious organic disease, mental illness, including any uncontrolled urinary, respiratory, circulation, nervous, digestive, endocrine, spirit, immune system diseases and tumor.
7. Suspected liver cancer or alpha feto protein (AFP) > 100ng/ml.
8. Neutrophil count < 2.5×109/L, or hemoglobin < 100g/L, or platelet < 80×109/L.
9. Pregnant or lactating women.
10. Allergic constitution, allergy history for blood products, known allergy to experimental drugs.
11. Alcohol or drug addiction, drug use history evidence within one year before enrolled in the study.
12. Received immunosuppressive or other immune modulators (including thymosin) or systemic cytotoxic drug 6 months before enrolled in the study.
13. Incompliance during antiviral therapy.
14. Enrolled in other clinical trials at present, and possible to be against the treatment and observation index.
15. Unable or unwilling to provide informed consent or fails to comply with the requirements of the study.
16. Other serious conditions that may hamper clinical trials.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-12 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
the rate of hepatitis B surface antigen (HBsAg) seroconversion | At week 48

SECONDARY OUTCOMES:
The rates of serum hepatitis B surface antigen (HBsAg) negative | At Baseline and at week 4, 12, 24, 36 and 48
the decreased levels of serum hepatitis B surface antigen (HBsAg) | At Baseline and at week 4, 12, 24, 36 and 48
Number of participants with adverse events as a measure of safety and tolerability | at baseline and up to week 48 week
The frequency of hepatitis B virus (HBV)-specific T cells | At baseline and at week 4, 12, 24, 36 and 48
The frequency of hepatitis B virus (HBV)-specific B cells | At baseline and at week 4, 12, 24, 36 and 48
liver hepatitis B surface antigen (HBsAg) levels | At baseline and week 48

OTHER OUTCOMES:
plasma hepatitis B virus (HBV) DNA load | At Entry and at Weeks 24 and 48
Hepatitis B virus (HBV) serum markers (HBsAg, HBsAb, HBeAg, HBeAb, HBcAb) | At baseline and at week 24 and 48

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Sheng Wang, M.D., Principal Investigator — Research Center for Biotherapy
Locations (1):
- Beijing 302 Hospital, Beijing, China

REFERENCES:
- [Background] Xu DZ, Wang XY, Shen XL, Gong GZ, Ren H, Guo LM, Sun AM, Xu M, Li LJ, Guo XH, Zhen Z, Wang HF, Gong HY, Xu C, Jiang N, Pan C, Gong ZJ, Zhang JM, Shang J, Xu J, Xie Q, Wu TF, Huang WX, Li YG, Xu J, Yuan ZH, Wang B, Zhao K, Wen YM; YIC Efficacy Trial Study Team. Results of a phase III clinical trial with an HBsAg-HBIG immunogenic complex therapeutic vaccine for chronic hepatitis B patients: experiences and findings. J Hepatol. 2013 Sep;59(3):450-6. doi: 10.1016/j.jhep.2013.05.003. Epub 2013 May 11. PMID 23669281
- [Background] Shouval D. Focus: quantitative HBsAg measurement as a new surrogate marker for assessment of hepatic fibrosis in HBeAg+ chronic hepatitis B. J Hepatol. 2013 Jun;58(6):1063-4. doi: 10.1016/j.jhep.2013.03.002. Epub 2013 Mar 14. No abstract available. PMID 23499728
- [Background] Seto WK, Wong DK, Fung J, Huang FY, Lai CL, Yuen MF. Reduction of hepatitis B surface antigen levels and hepatitis B surface antigen seroclearance in chronic hepatitis B patients receiving 10 years of nucleoside analogue therapy. Hepatology. 2013 Sep;58(3):923-31. doi: 10.1002/hep.26376. Epub 2013 Jul 24. PMID 23468172
- [Background] Tseng TC, Liu CJ, Yang HC, Su TH, Wang CC, Chen CL, Hsu CA, Kuo SF, Liu CH, Chen PJ, Chen DS, Kao JH. Serum hepatitis B surface antigen levels help predict disease progression in patients with low hepatitis B virus loads. Hepatology. 2013 Feb;57(2):441-50. doi: 10.1002/hep.26041. Epub 2012 Dec 6. PMID 22941922